CLINICAL TRIAL: NCT06584617
Title: A Prospective, 8-week, Multi-centre, Randomised, Open-label Clinical Investigation Comparing Clinical Efficacy and Safety of Berovenal® with a Reference Amorphous Hydrogel in Subjects with Shallow, Non-infected, Chronic Diabetic Foot Ulcer
Brief Title: The Purpose of This Study is to Assess Clinical Efficacy and Safety of Berovenal® Intended to Promote Treatment and to Expedite Chronic Diabetic Foot Ulcer Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VULM s.r.o. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BER202001
Record Dates: First submitted 2024-08-21; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Berovenal® (Experimental)
  Interventions: Device: Berovenal®
- NU-GEL Hydrogel with Alginate (Active Comparator)
  Interventions: Device: NU-GEL Hydrogel with Alginate

INTERVENTIONS:
Device: Berovenal® — Easy to spread, water-washable, light brown, turbid hydrogel in tube containing 30 g of hydrogel and closed with a plastic screw cap.
  Arms: Berovenal®
Device: NU-GEL Hydrogel with Alginate — Transparent, easy to spread and water-washable hydrogel in ampoule (concertina pack) containing 25 g or 15 g of hydrogel and closed with a plastic cap.
  Arms: NU-GEL Hydrogel with Alginate

SUMMARY:
The goal of this clinical investigation is to evaluate clinical efficacy of medical device Berovenal® intended to promote treatment and to expedite healing of chronic diabetic foot ulcer in male or female subjects aged 18-85 years with diabetes mellitus (type 1 or 2) and with present diabetic foot ulcer by providing moist environment similar to intracellular environment of the damaged tissue. It will also learn about the safety of medical device Berovenal®.

The main questions it aims to answer are:

* Does medical device Berovenal® lower the size of diabetic foot ulcer?
* What medical problems do participants have when using medical device Berovenal®?

Researchers will compare medical device Berovenal® to a reference device (device with similar purpose of use).

Participants will:

* Use medical device Berovenal® or a reference device every day for 8 weeks or to the time point when the diabetic foot is closed
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their symptoms and the number of times they use medical device Berovenal® or a reference device

ELIGIBILITY:
Inclusion Criteria:

* male, or female subjects aged 18-85 years;
* diabetes mellitus (type 1 or 2) documented at least 12 months prior to Visit 1;
* presence of a diabetic foot ulcer meeting the following criteria (Index ulcer):

  * grade 1 or 2 according to the Wagner classification;
  * if applicable, surgically debrided ≥ 7 days prior to Visit 1;
  * at the time of randomisation:
* sized 1 - 25 cm2;
* present for ≥ 14 days;
* offloaded for ≥ 7 days;
* not infected.
* HbA1c ≤ 10% (DCCT) or 85.8 mmol/mol (IFCC) at Visit 1;
* willing and able to comply with the scheduled procedures;
* legally capable, able to understand the provided information and willing to sign the informed consent form.

Exclusion Criteria:

* known contraindication for application of hydrogel dressings, incl. Berovenal® and NU-GEL Hydrogel with Alginate;
* at the time of randomisation - documented reduction in Index ulcer area by > 20%, as compared to its size at Visit 1;
* Index ulcer primarily caused by a medical condition other than diabetes mellitus;
* inadequate arterial circulation to the foot documented within 28 days prior to Visit 1, or during the screening period:

  * Ankle-brachial Index < 0.7 or > 1.3 and/or
  * Toe-brachial Index < 0.7;
* presence of acute Charcot's neuro-arthropathy, or osteomyelitis, on the affected foot within 3 months prior to Visit 1;
* use of wound dressings that include growth factors, bioengineered tissues, or skin substitutes within 14 days prior to Visit 1, or documented intention to use them during the subject's participation;
* use of any investigational drug(s) or device(s), systemic immunosuppressive treatment (including systemic corticosteroids), or application of topical steroids to the Index ulcer surface, within 28 days prior to Visit 1;
* use of cytotoxic chemotherapy and/or radiotherapy within 6 months prior to Visit 1;
* known history of bone cancer or metastatic disease of the affected limb;
* poor nutritional status;
* presence of an on-going uncontrolled renal, hepatic, cardiovascular or other disease that could pose an additional risk for the participant, or could significantly influence interpretation of the results (as evaluated by the investigator);
* known history of non-compliance and/or presence of any condition(s) seriously compromising the subject's ability to adhere to the procedures required by this Clinical Investigational Plan;
* pregnant or breast-feeding females;
* females of childbearing potential not using an effective method of contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical efficacy based on comparison of the percentage reduction in Index ulcer area. | 8 weeks

SECONDARY OUTCOMES:
Evaluation of clinical efficacy based on proportion of subjects who achieved complete closure of Index ulcers | 8 weeks
Evaluation of clinical efficacy based on median time until complete Index ulcer closure | 8 weeks
Evaluation of clinical efficacy based on proportion of subjects who achieved a reduction in the Index ulcer area by ≥ 80% | 4, 6 and 8 weeks
Evaluation of clinical efficacy based on mean percentage change of the Index ulcer area | 2, 4, 6 and 8 weeks
Evaluation of clinical efficacy based on improvement in the subject's reported quality of life assessed by the Wound-QoL | 2, 4, 6 and 8 weeks
Evaluation of safety based on proportion of target wounds with a documented wound infection | 8 weeks
Evaluation of safety occurrence of adverse events, device failures or complaints | 8 weeks
Evaluation of clinical efficacy based on wound healing process | 2, 4, 6 and 8 weeks
  The analysis will inolve evaluation wound depth, presence of granulation tissue, exsudate and infection at individual time points.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (2):
  - Klinik Kösching, Kösching, Eichstatt
  - Universitätsklinikum Heidelberg, Heidelberg
- Poland (7):
  - Diab Serwis Popenda Spółka Jawna, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - MIKOMED Sp. z o.o., Lodz
  - Wojewódzka Poradnia Diabetologiczna, Gabinet Stopy Cukrzycowej, Olsztyn
  - Centrum Medyczne Omedica Jarosław Opiela I Beata Opiela Spółka Jawna, Poznan
  - Ginemedica Sp. z o.o. Sp. k., Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided